CLINICAL TRIAL: NCT00848354
Title: A Randomized, Open-label Study In The Latin America Region Comparing The Safety And Efficacy Of Etanercept With Conventional Dmard Therapy In Subjects With Rheumatoid Arthritis.
Brief Title: Open-Label Study Comparing Etanercept to Conventional Disease Modifying Antirheumatic Drug (DMARD) Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-4532; B1801004 (Other: Alias Study Number)
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: enbrel; moderate arthritis; severe arthritis; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 Etanercept + methotrexate (Experimental): Phase 1: Etanercept + methotrexate
  Interventions: Biological: Phase 1: Etanercept; Drug: Phase 1: Methotrexate; Drug: Phase 2: Optional ETN, SSZ, HCQ, MTX
- Phase 1 Conventional DMARD (SSZ or HCQ) + MTX (Active Comparator): Phase 1: Sulfasalazine (SSZ) + methotrexate (MTX) OR Phase 1: Hydrocholoquine (HCQ) + methotrexate
  Interventions: Drug: Phase 1: Methotrexate; Drug: Phase 1: Conventiaonal DMARD

INTERVENTIONS:
Biological: Phase 1: Etanercept — Phase 1: prefilled syringe 50mg/ml, administered once weekly for study weeks 0 - 24
  Other Names: Enbrel
  Arms: Phase 1 Etanercept + methotrexate
Drug: Phase 1: Methotrexate — Phase 1: oral tablet, 2.5mg, dose variable from 7.5mg to 25mg, once weekly for study weeks 0 - 24.
  Arms: Phase 1 Etanercept + methotrexate
Drug: Phase 2: Optional ETN, SSZ, HCQ, MTX — Phase 2: All therapies are optional and may include any combination of the following: ETN, SSZ, HCQ, MTX Phase 2: Optional ETN: prefilled syringe 50mg/ml, dose variable after study week 24 to week 128.
  Phase 2: Optional SSZ: oral tablet, 0.5gm, dose variable per approved local label recommendations after study week 24 to week 128.
  Phase 2: HCQ: oral tablet, 200mg, dose variable per approved local label recommendations after study week 24 to week 128.
  Phase 2: MTX: oral tablet, 2.5mg dose variable after week 24 to week 128.
  Arms: Phase 1 Etanercept + methotrexate
Drug: Phase 1: Methotrexate — Phase 1: oral tablet, 2.5mg dose variable from 7.5mg to 25mg, once weekly for study weeks 0 - 24.
  Arms: Phase 1 Conventional DMARD (SSZ or HCQ) + MTX
Drug: Phase 1: Conventiaonal DMARD — Phase 1: SSZ: oral tablet, 0.5gm, dose variable per approved local label recommendations. OR Phase 1: HCQ: oral tablet, 200mg, dose variable per approved local label recommendations.
  Arms: Phase 1 Conventional DMARD (SSZ or HCQ) + MTX

SUMMARY:
The purpose of this 2 phased, open-label study is to compare the safety and efficacy of etanercept with conventional Disease Modifying Antirheumatic Drug (DMARD) therapy in Latin American subjects with moderate to severe rheumatoid arthritis over 128 weeks. Phase 1 is a randomized 24 week treatment period; Phase 2 is an optional open-label 104 week period that allows the investigator to choose continuation with the phase I treatment or the addition, discontinuation or titration of other DMARD therapy already being utilized for the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis (RA)
* Currently receiving a suboptimal response to a stable dose of methotrexate for treatment of Rheumatoid Arthritis (RA)
* Active Rheumatoid Arthritis (RA) at time of screening and baseline

Exclusion Criteria:

* Previous or current treatment with etanercept, other tumor necrosis factor-alpha inhibitors, or other biologic agents
* Concurrent treatment with a Disease Modifying Antirheumatic Drug (DMARD), other than methotrexate, at screening
* Receipt of any Disease Modifying Antirheumatic Drug (DMARD), other than methotrexate, within 3 months before screening

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Argentina (13):
  - Investigaciones Reumatológicas y Osteológicas, Buenos Aires, Argentina
  - OMI, Buenos Aires, Buenos Aires
  - Centro de Investigaciones en Enfermedades Reumaticas, Buenos Aires, Buenos Aires
  - Hospital Britanico, Buenos Aires, Buenos Aires
  - Atencion Integral en Reumatologia, Buenos Aires, Buenos Aires
  - Consultorios Especializados en Investigaciones Medicas, Capital Federal, Buenos Aires
  - Hospital Escuela Gral. San Martin, Corrientes, Corrientes Province
  - CER San Juan, San Juan, Provinica de San Juan
  - Instituto CAICI, Rosario, Santa Fe Province
  - Centro de Investigaciones Reumatologicas, San Miguel de Tucumán, Tucumán Province
  - Centro de Osteopatías Médicas, Buenos Aires
  - Sanatorio Mayo, Córdoba
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Chile (2):
  - Dr Miranda Private Practice, Santiago, Santiago Metropolitan
  - Hospital del Salvador, Santiago, Santiago Metropolitan
- Colombia (11):
  - Reumalab, Medellín, Antioquia
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - IPS Centro Integral de Rematología del Caribe S.A.S CIRCARIBE S.A.S Sede 1, Barranquilla, Atlántico
  - IPS Centro Integral de Rematología del Caribe S.A.S CIRCARIBE S.A.S Sede 2, Barranquilla, Atlántico
  - Centro Integral de Reumatologia e Inmunologia LTDA, Bogota, Cundinamarca
  - Foqus Ips Ltda, Bogota, Cundinamarca
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogota, Cundinamarca
  - Riesgo de fractura S.A. Clinica de Artritis y Rehabilitacion, Bogota, Cundinamarca
  - Preventive Care Ltda, Chía, Cundinamarca
  - Centro Medico Carlos Ardila Lulle, Bucaramanga, Santander Department
  - Servimed EU, Bucaramanga, Santander Department
- Mexico (5):
  - Centro de Investigación y Biomedicina de Chihuahua, Chihuahua City, Chihuahua
  - Hospital Christus Mugerza, Chihuahua City, Chihuahua
  - Hospital Christus Muguerza del Parque, Chihuahua City, Chihuahua
  - Hospital Angeles Chapalita, Guadajara, Jalisco
  - Centro de Especialidades Medicas del Sureste SA de CV, Mérida, Yucatán
- Panama (2):
  - Centro de Infusion Marbella, Panama City
  - Centro de Investigacion Marbella, Panama City

REFERENCES:
- [Derived] de la Vega M, Guerra Bautista G, Xavier RM, Pacheco-Tena C, Solano G, Pedersen RD, Szumski AE, Borlenghi C, Santana K, Vlahos B. Predictors of response to etanercept-methotrexate treatment: a post hoc logistic regression analysis of a randomized, open-label study in Latin American patients with rheumatoid arthritis. Adv Rheumatol. 2021 Sep 8;61(1):56. doi: 10.1186/s42358-021-00213-4. PMID 34496979
- [Derived] Guerra Bautista G, Xavier RM, de la Vega M, Simon-Campos JA, Solano G, Pedersen RD, Vlahos B, Borlenghi C. Clinical Improvements as Predictors of Improvements in Patient-Reported Outcomes: Post Hoc Analysis of a Randomized, Open-Label Study of Etanercept in Latin American Patients with Rheumatoid Arthritis. Open Access Rheumatol. 2019 Dec 12;11:275-281. doi: 10.2147/OARRR.S228866. eCollection 2019. PMID 31849542
- [Derived] Machado DA, Guzman R, Xavier RM, Simon JA, Mele L, Shen Q, Pedersen R, Kotak S, Vlahos B. Two-Year Safety and Efficacy Experience in Patients with Methotrexate-Resistant Active Rheumatoid Arthritis Treated with Etanercept and Conventional Disease-Modifying Anti-rheumatic Drugs in the Latin American Region. Open Rheumatol J. 2016 Feb 29;10:13-25. doi: 10.2174/1874312901610010013. eCollection 2016. PMID 27006728
- [Derived] Fleischmann R, Koenig AS, Szumski A, Nab HW, Marshall L, Bananis E. Short-term efficacy of etanercept plus methotrexate vs combinations of disease-modifying anti-rheumatic drugs with methotrexate in established rheumatoid arthritis. Rheumatology (Oxford). 2014 Nov;53(11):1984-93. doi: 10.1093/rheumatology/keu235. Epub 2014 Jun 6. PMID 24907147
- [Derived] Machado DA, Guzman RM, Xavier RM, Simon JA, Mele L, Pedersen R, Ferdousi T, Koenig AS, Kotak S, Vlahos B. Open-label observation of addition of etanercept versus a conventional disease-modifying antirheumatic drug in subjects with active rheumatoid arthritis despite methotrexate therapy in the Latin American region. J Clin Rheumatol. 2014 Jan;20(1):25-33. doi: 10.1097/RHU.0000000000000055. PMID 24356474
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-4532&StudyName=Open-Label%20Study%20Comparing%20Etanercept%20to%20Conventional%20Disease%20Modifying%20Antirheumatic%20Drug%20%28DMARD%29%20Therapy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 3 periods - Phase 1 (week 0-week 24), Phase 2 Year 1 (week 24-week 76), and Phase 2 Year 2 (week 76-week 128). 429 participants were randomly assigned to open label etanercept + methotrexate or open label conventional disease-modifying antirheumatic drug (DMARD) + methotrexate in a 2:1 allocation, respectively.
Pre-assignment Details: Five participants (etanercept + methotrexate: 3, DMARD + methotrexate: 2) were randomized but did not receive study treatment. These participants were either randomized in error or withdrew consent before receiving the first dose. Phase 1 DMARD therapy was either hydroxychloroquine (HCQ) or sulfsalazine (SSZ), as selected by the investigator.
Groups:
- Etanercept + Methotrexate: Phase 1: Etanercept 50 mg injection subcutaneously (s.c.) once weekly along with methotrexate tablet (7.5-25 mg) orally once weekly either in single dose or in 2 divided doses for 24 weeks. Phase 2: During the optional Phase 2-period (week 24-week 128), the participants could remain on etanercept and methotrexate, or a non-biologic DMARD the investigator preferred in accordance with the local label (SSZ or HCQ) could be added in exchange for or in addition to etanercept. Methotrexate could be continued, discontinued or titrated. Phase 1 reporting groups were used also for Phase 2 data, regardless of the participant's Phase 2 treament regimen.
- DMARD + Methotrexate: Phase 1: Conventional DMARD combination therapy (SSZ or HCQ) tablets administered as per local prescribing practice, along with methotrexate tablet (7.5-25 mg) orally once weekly either in single dose or in 2 divided doses for 24 weeks. Phase 2: During the optional Phase 2-period (week 24-week 128), the participants could remain on DMARD (SSZ or HCQ) and methotrexate, or a DMARD the investigator preferred in accordance with the local label (HCQ, SSZ, and/or etanercept) could be added in exchange for or in addition to the Phase 1 DMARD (SSZ or HCQ). Methotrexate and the DMARD administered in Phase 1 could be continued, discontinued or titrated. Phase 1 reporting groups were used also for Phase 2 data, regardless of the participant's Phase 2 treament regimen.
Period: Phase 1
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Started | 281 (One participant was randomized to the Etanercept + Methotrexate group but received SSZ in error.) | 143
Completed | 269 | 129
Not Completed | 12 | 14
Not completed — Adverse Event | 5 | 4
Not completed — Discontinuation of study by sponsor | 2 | 1
Not completed — Failed to return | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Unspecified Reason | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lack of Efficacy | 0 | 1
Period: Phase 2 Year 1
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Started | 260 (Randomized Phase 1 treatment assignment. 9 participants discontinued between Phase 1 and Phase 2.) | 126 (Randomized Phase 1 treatment assignment. 3 participants discontinued between Phase 1 and Phase 2.)
Completed | 242 | 120
Not Completed | 18 | 6
Not completed — Adverse Event | 7 | 2
Not completed — Death | 1 | 0
Not completed — Failed to Return | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Unspecified Reason | 3 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Subject Request | 1 | 2
Period: Phase 2 Year 2
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Started | 241 (Randomized Phase 1 treatment assignment. 1 participant discontinued between Year 1 and Year 2.) | 120 (Randomized Phase 1 treatment assignment.)
Completed | 218 | 113
Not Completed | 23 | 7
Not completed — Adverse Event | 12 | 2
Not completed — Death | 2 | 0
Not completed — Failed to return | 3 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Unspecified Reason | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Subject Request | 1 | 1
Not completed — Unsatisfactory Response - Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participant with documented use of at least 1 dose of test article - Baseline characteristics from Phase 1 CSR are provided.
Groups:
- Etanercept + Methotrexate: Phase 1: Etanercept 50 mg injection s.c. once weekly along with methotrexate tablet (7.5-25 mg) orally once weekly either in single dose or in 2 divided doses for 24 weeks. Phase 2: During the optional Phase 2-period (week 24-week 128), the participants could remain on etanercept and methotrexate, or a non-biologic DMARD the investigator preferred in accordance with the local label (SSZ or HCQ) could be added in exchange for or in addition to etanercept. Methotrexate could be continued, discontinued or titrated. Phase 1 reporting groups were used also for Phase 2 data, regardless of the participant's Phase 2 treament regimen.
- Total: Total of all reporting groups
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate | Total
Number analyzed (Participants) | 281 | 143 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.99) | 48.7 (11.40) | 48.5 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 129 | 377
  Male | 33 | 14 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 (ACR50) Response at Week 24
Description: ACR50 response: greater than or equal to 50 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 50 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of the Health Assessment Questionnaire; HAQ); and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: Modified intent-to-treat (mITT) population included all participants who took at least 1 dose of study drug and had at least 1 post-randomization visit that included evaluation of tender and swollen joints and at least 3 of other 5 variables required to calculate ACR50. Last Observation carried forward (LOCF) method was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
Percentage of participants | 62.01 | 23.24
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Cochran-Mantel-Haenszel chi-square test, stratified by country, was used to calculate p-value. Assuming ACR50 response at Week 24 to be 23% in the DMARD combination therapy group and 37% in the etanercept + methotrexate group, a study enrolling 276 participants assigned to etanercept + methotrexate and 138 participants assigned to DMARD combination therapy has 80% power to reject the null hypothesis of no difference in response rates testing at the type I error = 0.05 level; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

2. Secondary Outcome: Change From Baseline in HAQ Score at Week 24
Description: HAQ: self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ score range: 0-3: without any difficulty: 0, with some difficulty: 1, with much difficulty: 2, unable to do: 3. HAQ total scores expressed as overall mean score with range 0-3: 0-0.25: normal functioning; 0.25-0.5: mild functional limitation; 0.5-1: moderate functional limitation; more than 1: significant functional limitation.
Time Frame: Baseline and Week 24
Population: mITT population included all participants who took at least 1 dose of study drug and had at least 1 post-randomization visit that included evaluation of tender and swollen joints and at least 3 of other 5 variables required to calculate ACR50. LOCF method was used.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 141
Units on a scale
  Baseline | 1.55 (0.05) | 1.51 (0.07)
  Change at Week 24 | -0.85 (0.04) | -0.51 (0.06)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Analysis of covariance (ANCOVA) model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

3. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Score at Week 24
Description: The SF-36 is standardized 36-item survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health perception, vitality, and mental health. Domain scores range from 0-100, with greater scores reflecting better health status. Two additional overall summary scores - physical and mental component scores - were also obtained. Summary scores are standardized where the general population mean is 50 with a standard deviation of 10. Greater scores again indicate better health status.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 278 | 141
Units on a scale
  Baseline, Vitality domain | 12.46 (0.28) | 12.39 (0.36)
  Baseline, Mental component | 40.50 (0.78) | 40.41 (1.00)
  Baseline, Physical component | 30.42 (0.50) | 30.18 (0.64)
  Change at Week 24, Vitality domain | 3.79 (0.27) | 2.36 (0.35)
  Change at Week 24, Mental component | 7.33 (0.73) | 3.32 (0.95)
  Change at Week 24, Physical component | 12.44 (0.65) | 7.36 (0.84)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for vitality domain at Week 24; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for mental component at Week 24; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for physical component at Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

4. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Total Sharp Score (vdH mTSS), Annualized, at Week 24
Description: mTSS: sum of erosion and joint space narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Each x-ray visit included 4 films, each of which were read by 2 readers. The mTSS was calculated by the images scored for erosions and JSN. An increase in mTSS from Baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Week 24
Population: Radiographic intent-to-treat (xITT) population included all participants who took at least 1 dose of study drug and had evaluable radiographic data at Baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 247 | 119
units on a scale
  Baseline | 31.19 (4.06) | 46.35 (5.35)
  Week 24 | 0.40 (0.36) | 1.37 (0.47)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model on ranks of change in mTSS with treatment group and center main effects and the Baseline rank as covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0270, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

5. Secondary Outcome: Change From Baseline in Disease Activity Score Based on a 28-joint Count (DAS28) at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS28 calculated from the number of swollen joints and painful joints using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour; mm/hour) and the participant's general health using a 100 mm-visual analog scale (VAS). DAS28<3.2 indicates low disease activity and DAS28<2.6 remission.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 2 (N: 275, 139) | -1.50 (0.07) | -0.67 (0.09)
  Week 4 (N: 278, 142) | -2.15 (0.08) | -1.27 (0.10)
  Week 8 (N: 279, 142) | -2.59 (0.09) | -1.54 (0.11)
  Week 12 (N: 279, 142) | -2.82 (0.09) | -1.83 (0.12)
  Week 16 (N: 279, 142) | -3.01 (0.09) | -1.84 (0.12)
  Week 20 (N: 279, 142) | -3.15 (0.09) | -1.84 (0.12)
  Week 24 (N: 279, 142) | -3.20 (0.09) | -1.70 (0.12)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-values. ANCOVA was ran at each time-point shown, however as p-values obtained were identical, only one p-value is presented (which is applicable to each time-point - Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24 - independently); Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

6. Secondary Outcome: Change From Baseline in DAS28 at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: DAS28 calculated from the number of swollen joints and painful joints using the 28 joints count, the ESR (mm/hour) and the participant's general health using a 100 mm-VAS. DAS28<3.2 indicates low disease activity and DAS28<2.6 remission.
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: mITT population (LOCF) was used. Phase 2 Year 1 (week 37-week 76)-sample size (Etanercept + Methotrexate, DMARD + Methotrexate: 260, 126) is different from Phase 2 Year 2 (week 89-week 128)-sample size (241, 120).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 37 (N: 260, 126) | -3.39 (1.34) | -3.08 (1.29)
  Week 50 (N: 260, 126) | -3.42 (1.32) | -3.33 (1.18)
  Week 63 (N: 260, 126) | -3.41 (1.31) | -3.42 (1.16)
  Week 76 (N: 260, 126) | -3.38 (1.33) | -3.36 (1.27)
  Week 89 (N: 241, 120) | -3.53 (1.34) | -3.47 (1.34)
  Week 102 (N: 241, 120) | -3.43 (1.26) | -3.47 (1.29)
  Week 115 (N: 241, 120) | -3.47 (1.31) | -3.28 (1.37)
  Week 128 (N: 241, 120) | -3.41 (1.40) | -3.51 (1.29)

7. Secondary Outcome: Summary of Changes in Therapy at the Beginning of Phase 2
Description: The investigators were allowed to alter each participant's therapy at the beginning of Phase 2. Continuations, discontinuations and additions made to Phase 1 treatment regimen were summarized.
Time Frame: Week 24
Population: mITT population included all participants who took at least 1 dose of study drug and had at least 1 post-randomization visit that included evaluation of tender and swollen joints and at least 3 of other 5 variables required to calculate ACR50. LOCF method was used. One participant was randomized to etanercept but received SSZ in Phase 1.
Measure: Number; unit: participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
participants
  No change: Etanercept | 259 | NA — Participants did not receive etanercept during Phase 1.
  No change: HCQ | NA — Participants did not receive HCQ during Phase 1. | 29
  No change: Methotrexate | 260 | 126
  No change: SSZ | NA — Participants did not receive SSZ during Phase 1. | 11
  Added Etanercept | 1 | 105
  Added HCQ | 8 | NA — Participants already received HCQ during Phase 1.
  Added SSZ | 3 | NA — Participants already received SSZ during Phase 1.
  Discontinued HCQ | NA — Participants did not receive HCQ during Phase 1. | 35
  Discontinued SSZ | 1 | 51

8. Secondary Outcome: Percentage of Participants Achieving ACR50 Response at Week 2, Week 4, Week 8, Week 12, Week 16, and Week 20
Description: ACR50 response: greater than or equal to 50 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 50 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, and Week 20
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 278, 140) | 15.83 | 2.86
  Week 4 (N: 279, 142) | 31.54 | 8.45
  Week 8 (N: 279, 142) | 42.29 | 16.90
  Week 12 (N: 279, 142) | 52.33 | 21.13
  Week 16 (N: 279, 142) | 56.27 | 24.65
  Week 20 (N: 279, 142) | 59.14 | 27.46
  Week 24 (N: 279, 142) | 62.01 | 23.24
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.39, 95% CI 2-sided [2.25 to 18.2]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.99, 95% CI 2-sided [2.62 to 9.49]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.6, 95% CI 2-sided [2.19 to 5.94]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.10, 95% CI 2-sided [2.57 to 6.53]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.93, 95% CI 2-sided [2.51 to 6.16]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.82, 95% CI 2-sided [2.46 to 5.93]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.39, 95% CI 2-sided [3.41 to 8.53]

9. Secondary Outcome: Percentage of Participants Achieving ACR50 Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: ACR50 response: greater than or equal to 50 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 50 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of HAQ); and ESR.
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 67.31 | 53.17
  Week 50 (N: 260, 126) | 65.77 | 60.32
  Week 63 (N: 260, 126) | 68.46 | 62.70
  Week 76 (N: 260, 126) | 67.31 | 58.73
  Week 89 (N: 241, 120) | 73.44 | 60.83
  Week 102 (N: 241, 120) | 73.44 | 61.67
  Week 115 (N: 241, 120) | 72.61 | 59.17
  Week 128 (N: 241, 120) | 70.54 | 65.00

10. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: ACR20 response: greater than or equal to 20 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 20 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 278, 140) | 47.84 | 19.29
  Week 4 (N: 279, 142) | 63.80 | 34.51
  Week 8 (N: 279, 142) | 73.84 | 49.30
  Week 12 (N: 279, 142) | 79.57 | 54.93
  Week 16 (N: 279, 142) | 84.23 | 57.75
  Week 20 (N: 279, 142) | 84.59 | 58.45
  Week 24 (N: 279, 142) | 83.15 | 50.00
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.84, 95% CI 2-sided [2.37 to 6.21]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.34, 95% CI 2-sided [2.19 to 5.11]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.90 to 4.43]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.20, 95% CI 2-sided [2.06 to 4.96]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.91, 95% CI 2-sided [2.46 to 6.21]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.90, 95% CI 2-sided [2.45 to 6.22]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.94, 95% CI 2-sided [3.13 to 7.78]

11. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: ACR20 response: greater than or equal to 20 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 20 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of HAQ); and ESR.
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 86.92 | 80.95
  Week 50 (N: 260, 126) | 90.00 | 86.51
  Week 63 (N: 260, 126) | 88.85 | 91.27
  Week 76 (N: 260, 126) | 89.23 | 87.30
  Week 89 (N: 241, 120) | 90.87 | 89.17
  Week 102 (N: 241, 120) | 91.70 | 90.83
  Week 115 (N: 241, 120) | 90.04 | 83.33
  Week 128 (N: 241, 120) | 89.21 | 89.17

12. Secondary Outcome: Percentage of Participants Achieving ACR70 Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: ACR70 response: greater than or equal to 50 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 70 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 278, 140) | 3.60 | 0.71
  Week 4 (N: 279, 142) | 7.17 | 2.11
  Week 8 (N: 279, 142) | 16.13 | 3.52
  Week 12 (N: 279, 142) | 20.07 | 4.23
  Week 16 (N: 279, 142) | 27.60 | 9.15
  Week 20 (N: 279, 142) | 30.11 | 10.56
  Week 24 (N: 279, 142) | 34.77 | 11.27
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p = 0.1086, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.19, 95% CI 2-sided [0.66 to 40.9]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p = 0.0392, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.58, 95% CI 2-sided [1.04 to 12.3]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.27, 95% CI 2-sided [2.04 to 13.6]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.69, 95% CI 2-sided [2.39 to 13.6]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.78, 95% CI 2-sided [2.02 to 7.09]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.65, 95% CI 2-sided [2.02 to 6.60]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.20, 95% CI 2-sided [2.36 to 7.46]

13. Secondary Outcome: Percentage of Participants Achieving ACR70 Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: ACR70 response: greater than or equal to 70 percent improvement from Baseline in tender joint count and swollen joint count; and greater than or equal to 70 percent improvement from Baseline in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; participant's self-assessed disability (disability index of HAQ); and ESR.
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 40.38 | 30.16
  Week 50 (N: 260, 126) | 45.00 | 32.54
  Week 63 (N: 260, 126) | 39.62 | 34.13
  Week 76 (N: 260, 126) | 41.92 | 34.13
  Week 89 (N: 241, 120) | 53.11 | 38.33
  Week 102 (N: 241, 120) | 48.96 | 36.67
  Week 115 (N: 241, 120) | 48.55 | 35.00
  Week 128 (N: 241, 120) | 48.96 | 40.00

14. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS calculated from number of painful joints using the ritchie articular index (RAI), number of swollen joints using the same 44 joints as in RAI, ESR (mm/hour) and participant's general health using a 100 mm-VAS. DAS≤2.4 indicates low disease activity and DAS<1.6 remission.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 2 (N: 274, 139) | -1.42 (0.07) | -0.65 (0.09)
  Week 4 (N: 277, 142) | -2.07 (0.07) | -1.29 (0.09)
  Week 8 (N: 278, 142) | -2.45 (0.07) | -1.55 (0.10)
  Week 12 (N: 278, 142) | -2.67 (0.08) | -1.79 (0.10)
  Week 16 (N: 278, 142) | -2.82 (0.08) | -1.86 (0.10)
  Week 20 (N: 278, 142) | -2.95 (0.08) | -1.85 (0.10)
  Week 24 (N: 278, 142) | -2.97 (0.08) | -1.72 (0.10)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

15. Secondary Outcome: Change From Baseline in DAS at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: DAS calculated from number of painful joints using RAI, number of swollen joints using the same 44 joints as in RAI, ESR (mm/hour) and participant's general health using a 100 mm-VAS. DAS≤2.4 indicates low disease activity and DAS<1.6 remission.
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 37 (N: 259, 126) | -3.13 (1.28) | -2.94 (1.25)
  Week 50 (N: 259, 126) | -3.21 (1.24) | -3.19 (1.12)
  Week 63 (N: 259, 126) | -3.17 (1.19) | -3.26 (1.19)
  Week 76 (N: 259, 126) | -3.18 (1.28) | -3.24 (1.23)
  Week 89 (N: 239, 120) | -3.29 (1.27) | -3.26 (1.38)
  Week 102 (N: 239, 120) | -3.24 (1.23) | -3.31 (1.31)
  Week 115 (N: 239, 120) | -3.28 (1.22) | -3.18 (1.41)
  Week 128 (N: 239, 120) | -3.23 (1.32) | -3.35 (1.38)

16. Secondary Outcome: Percentage of Participants Achieving DAS<2.4 (Low Disease Activity) Response at Week 24
Description: DAS calculated from number of painful joints using RAI, number of swollen joints using the same 44 joints as in RAI, ESR (mm/hour) and participant's general health using a 100 mm-VAS. DAS<2.4: low disease activity, DAS<1.6: remission.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 278 | 142
percentage of participants | 61.51 | 20.42
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.23, 95% CI 2-sided [3.88 to 10.00]

17. Secondary Outcome: Percentage of Participants Achieving DAS<1.6 (Remission) Response at Week 24
Description: as for outcome 16
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 278 | 142
percentage of participants | 28.78 | 4.93
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.79, 95% CI 2-sided [3.49 to 17.39]

18. Secondary Outcome: Percentage of Participants Achieving DAS Improvement of ≥0.6 From Baseline at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: as for outcome 16
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 274, 139) | 79.93 | 53.24
  Week 4 (N: 277, 142) | 90.97 | 66.90
  Week 8 (N: 278, 142) | 95.68 | 78.87
  Week 12 (N: 278, 142) | 95.32 | 81.69
  Week 16 (N: 278, 142) | 96.76 | 83.10
  Week 20 (N: 278, 142) | 97.12 | 83.10
  Week 24 (N: 278, 142) | 96.04 | 76.06
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.50, 95% CI 2-sided [2.24 to 5.46]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.99, 95% CI 2-sided [2.91 to 8.55]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.94, 95% CI 2-sided [2.93 to 12.02]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.57, 95% CI 2-sided [2.27 to 9.21]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.08, 95% CI 2-sided [2.74 to 13.48]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.86, 95% CI 2-sided [3.00 to 15.72]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.64, 95% CI 2-sided [3.74 to 15.63]

19. Secondary Outcome: Percentage of Participants Achieving DAS Improvement of ≥0.6 From Baseline at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 16
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 259, 126) | 98.07 | 96.83
  Week 50 (N: 259, 126) | 98.46 | 98.41
  Week 63 (N: 259, 126) | 96.91 | 99.21
  Week 76 (N: 259, 126) | 96.53 | 98.41
  Week 89 (N: 239, 120) | 97.49 | 98.33
  Week 102 (N: 239, 120) | 98.74 | 98.33
  Week 115 (N: 239, 120) | 98.33 | 96.67
  Week 128 (N: 239, 120) | 97.07 | 99.17

20. Secondary Outcome: Percentage of Participants Achieving DAS Improvement of ≥1.2 From Baseline at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: as for outcome 16
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 274, 139) | 57.66 | 30.22
  Week 4 (N: 277, 142) | 78.34 | 45.07
  Week 8 (N: 278, 142) | 84.89 | 58.45
  Week 12 (N: 278, 142) | 87.77 | 64.79
  Week 16 (N: 278, 142) | 92.09 | 67.61
  Week 20 (N: 278, 142) | 91.73 | 66.90
  Week 24 (N: 278, 142) | 91.01 | 60.56
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.15, 95% CI 2-sided [2.04 to 4.86]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.41, 95% CI 2-sided [2.85 to 6.82]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.99, 95% CI 2-sided [2.50 to 6.38]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.90, 95% CI 2-sided [2.37 to 6.41]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.58, 95% CI 2-sided [3.19 to 9.76]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.49, 95% CI 2-sided [3.16 to 9.52]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.59, 95% CI 2-sided [3.87 to 11.21]

21. Secondary Outcome: Percentage of Participants Achieving DAS Improvement of ≥1.2 From Baseline at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 16
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 259, 126) | 95.37 | 89.68
  Week 50 (N: 259, 126) | 96.53 | 96.03
  Week 63 (N: 259, 126) | 95.75 | 95.24
  Week 76 (N: 259, 126) | 94.21 | 96.03
  Week 89 (N: 239, 120) | 94.56 | 94.17
  Week 102 (N: 239, 120) | 95.40 | 97.50
  Week 115 (N: 239, 120) | 97.49 | 94.17
  Week 128 (N: 239, 120) | 94.14 | 95.83

22. Secondary Outcome: Percentage of Participants Achieving Moderate/Good DAS-Based European League Against Rheumatism (EULAR) Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from Baseline and the level of disease activity reached. Moderate or good DAS-based EULAR response was defined as:
  * DAS-value ≤3.7 and DAS-improvement from Baseline >0.6
  * DAS-value >3.7 and DAS-improvement from Baseline >1.2
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 274, 139) | 66.42 | 35.97
  Week 4 (N: 277, 142) | 84.12 | 52.11
  Week 8 (N: 278, 142) | 89.93 | 64.08
  Week 12 (N: 278, 142) | 91.01 | 69.72
  Week 16 (N: 278, 142) | 93.88 | 72.54
  Week 20 (N: 278, 142) | 94.6 | 73.94
  Week 24 (N: 278, 142) | 92.45 | 65.49
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.52, 95% CI 2-sided [2.30 to 5.40]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.87, 95% CI 2-sided [3.07 to 7.71]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.00, 95% CI 2-sided [2.98 to 8.41]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.55 to 7.58]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.81, 95% CI 2-sided [3.15 to 10.74]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.18, 95% CI 2-sided [3.25 to 11.73]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.45, 95% CI 2-sided [3.67 to 11.33]

23. Secondary Outcome: Percentage of Participants Achieving Moderate/Good Disease DAS-Based EULAR Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 22
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 259, 126) | 97.3 | 93.65
  Week 50 (N: 259, 126) | 97.3 | 97.62
  Week 63 (N: 259, 126) | 96.53 | 98.41
  Week 76 (N: 259, 126) | 95.37 | 97.62
  Week 89 (N: 239, 120) | 97.07 | 97.50
  Week 102 (N: 239, 120) | 97.49 | 97.50
  Week 115 (N: 239, 120) | 98.33 | 96.67
  Week 128 (N: 239, 120) | 96.23 | 98.33

24. Secondary Outcome: Percentage of Participants Achieving Good DAS-Based EULAR Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from Baseline and the level of disease activity reached. Good DAS-based EULAR response was defined as: DAS-value ≤2.4 and DAS-improvement from Baseline >1.2.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 274, 139) | 8.39 | 2.88
  Week 4 (N: 277, 142) | 24.55 | 7.75
  Week 8 (N: 278, 142) | 39.21 | 15.49
  Week 12 (N: 278, 142) | 48.2 | 22.54
  Week 16 (N: 278, 142) | 56.12 | 22.54
  Week 20 (N: 278, 142) | 58.99 | 24.65
  Week 24 (N: 278, 142) | 61.15 | 20.42
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p = 0.0349, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.09, 95% CI 2-sided [1.05 to 9.13]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.87, 95% CI 2-sided [1.98 to 7.60]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.52, 95% CI 2-sided [2.10 to 5.88]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.20, 95% CI 2-sided [2.02 to 5.06]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.78 to 6.96]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.80 to 6.90]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.13, 95% CI 2-sided [3.82 to 9.85]

25. Secondary Outcome: Percentage of Participants Achieving Good DAS-Based EULAR Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 24
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 259, 126) | 73.36 | 56.35
  Week 50 (N: 259, 126) | 72.2 | 69.05
  Week 63 (N: 259, 126) | 72.97 | 70.63
  Week 76 (N: 259, 126) | 73.75 | 64.29
  Week 89 (N: 239, 120) | 76.57 | 68.33
  Week 102 (N: 239, 120) | 77.41 | 70.83
  Week 115 (N: 239, 120) | 76.57 | 66.67
  Week 128 (N: 239, 120) | 75.73 | 70.00

26. Secondary Outcome: Percentage of Participants Achieving Moderate/Good DAS28-Based EULAR Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from Baseline and the level of disease activity reached. Moderate or good DAS28-based EULAR response was defined as:
  * DAS28-value ≤5.1 and DAS28-improvement from Baseline >0.6
  * DAS28-value >5.1 and DAS28-improvement from Baseline >1.2
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 275, 139) | 64 | 29.5
  Week 4 (N: 278, 142) | 81.29 | 48.59
  Week 8 (N: 279, 142) | 88.89 | 60.56
  Week 12 (N: 279, 142) | 91.4 | 64.79
  Week 16 (N: 279, 142) | 93.91 | 68.31
  Week 20 (N: 279, 142) | 94.62 | 67.61
  Week 24 (N: 279, 142) | 91.76 | 64.79
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.25, 95% CI 2-sided [2.74 to 6.60]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.60, 95% CI 2-sided [2.94 to 7.18]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.21, 95% CI 2-sided [3.15 to 8.61]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.77, 95% CI 2-sided [3.36 to 9.93]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.15, 95% CI 2-sided [3.91 to 13.09]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 8.43, 95% CI 2-sided [4.50 to 15.80]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.05, 95% CI 2-sided [3.50 to 10.47]

27. Secondary Outcome: Percentage of Participants Achieving Moderate/Good DAS28-Based EULAR Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 26
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 95.77 | 93.65
  Week 50 (N: 260, 126) | 96.15 | 95.24
  Week 63 (N: 260, 126) | 96.15 | 96.83
  Week 76 (N: 260, 126) | 95 | 96.83
  Week 89 (N: 241, 120) | 95.85 | 96.67
  Week 102 (N: 241, 120) | 95.02 | 96.67
  Week 115 (N: 241, 120) | 95.44 | 93.33
  Week 128 (N: 241, 120) | 92.95 | 97.50

28. Secondary Outcome: Percentage of Participants Achieving Good DAS28-Based EULAR Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from Baseline and the level of disease activity reached. Good DAS28-based EULAR response was defined as: DAS28-value ≤3.2 and DAS28-improvement from Baseline >1.2.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 275, 139) | 5.09 | 0.72
  Week 4 (N: 278, 142) | 10.79 | 4.93
  Week 8 (N: 279, 142) | 22.22 | 9.15
  Week 12 (N: 279, 142) | 30.11 | 12.68
  Week 16 (N: 279, 142) | 38.35 | 16.9
  Week 20 (N: 279, 142) | 43.01 | 15.49
  Week 24 (N: 279, 142) | 46.95 | 11.97
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p = 0.0250, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.40, 95% CI 2-sided [0.96 to 56.88]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p = 0.0466, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.00 to 5.45]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p = 0.0007, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.50 to 5.36]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.97, 95% CI 2-sided [1.70 to 5.18]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.85 to 5.05]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.12, 95% CI 2-sided [2.47 to 6.87]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.51, 95% CI 2-sided [3.72 to 11.38]

29. Secondary Outcome: Percentage of Participants Achieving Good DAS28-Based EULAR Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 28
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 53.08 | 37.3
  Week 50 (N: 260, 126) | 54.62 | 45.24
  Week 63 (N: 260, 126) | 55.38 | 50.79
  Week 76 (N: 260, 126) | 56.92 | 44.44
  Week 89 (N: 241, 120) | 60.58 | 50.83
  Week 102 (N: 241, 120) | 56.43 | 50.00
  Week 115 (N: 241, 120) | 56.85 | 45.83
  Week 128 (N: 241, 120) | 57.68 | 55.00

30. Secondary Outcome: Percentage of Participants Achieving DAS28<2.6 (Remission) Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: DAS28 calculated from number of swollen joints and painful joints using the 28 joints count, ESR (mm/hour) and participant's general health using a 100 mm-VAS. DAS28<3.2: low disease activity, DAS28<2.6: remission.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 275, 139) | 1.45 | 0
  Week 4 (N: 278, 142) | 4.32 | 2.11
  Week 8 (N: 279, 142) | 10.04 | 4.23
  Week 12 (N: 279, 142) | 14.7 | 5.63
  Week 16 (N: 279, 142) | 20.43 | 5.63
  Week 20 (N: 279, 142) | 28.67 | 6.34
  Week 24 (N: 279, 142) | 25.09 | 3.52
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p = 0.3054, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p = 0.4044, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.09, 95% CI 2-sided [0.58 to 7.53]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p = 0.0388, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.02 to 6.26]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p = 0.0059, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.89, 95% CI 2-sided [1.31 to 6.34]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.30, 95% CI 2-sided [1.99 to 9.29]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.94, 95% CI 2-sided [2.88 to 12.24]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 9.18, 95% CI 2-sided [3.61 to 23.32]

31. Secondary Outcome: Percentage of Participants Achieving DAS28<2.6 (Remission) Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 30
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 33.85 | 22.22
  Week 50 (N: 260, 126) | 36.54 | 26.19
  Week 63 (N: 260, 126) | 38.46 | 26.19
  Week 76 (N: 260, 126) | 33.46 | 23.02
  Week 89 (N: 241, 120) | 45.64 | 34.17
  Week 102 (N: 241, 120) | 36.93 | 36.67
  Week 115 (N: 241, 120) | 39.42 | 30.00
  Week 128 (N: 241, 120) | 39.83 | 33.33

32. Secondary Outcome: Percentage of Participants Achieving DAS28<3.2 (Low Disease Activity) Response at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: as for outcome 30
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 275, 139) | 5.09 | 0.72
  Week 4 (N: 278, 142) | 10.79 | 4.93
  Week 8 (N: 279, 142) | 22.22 | 9.15
  Week 12 (N: 279, 142) | 30.11 | 12.68
  Week 16 (N: 279, 142) | 38.35 | 16.9
  Week 20 (N: 279, 142) | 43.01 | 15.49
  Week 24 (N: 279, 142) | 46.95 | 11.97
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p = 0.0250, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.40, 95% CI 2-sided [0.96 to 56.88]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p = 0.0466, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.00 to 5.45]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p = 0.0007, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.50 to 5.36]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 2.97, 95% CI 2-sided [1.70 to 5.18]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.85 to 5.05]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.12, 95% CI 2-sided [2.47 to 6.87]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.51, 95% CI 2-sided [3.72 to 11.38]

33. Secondary Outcome: Percentage of Participants Achieving DAS28<3.2 (Low Disease Activity) Response at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 30
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 53.08 | 37.3
  Week 50 (N: 260, 126) | 54.62 | 45.24
  Week 63 (N: 260, 126) | 55.38 | 50.79
  Week 76 (N: 260, 126) | 56.92 | 44.44
  Week 89 (N: 241, 120) | 60.58 | 50.83
  Week 102 (N: 241, 120) | 56.43 | 50.00
  Week 115 (N: 241, 120) | 56.85 | 45.83
  Week 128 (N: 241, 120) | 57.68 | 55.00

34. Secondary Outcome: Percentage of Participants Achieving DAS28 Improvement of ≥0.6 From Baseline at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: as for outcome 30
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 275, 139) | 80.36 | 47.48
  Week 4 (N: 278, 142) | 89.93 | 69.01
  Week 8 (N: 279, 142) | 93.91 | 74.65
  Week 12 (N: 279, 142) | 95.34 | 79.58
  Week 16 (N: 279, 142) | 96.06 | 78.87
  Week 20 (N: 279, 142) | 96.77 | 78.17
  Week 24 (N: 279, 142) | 95.70 | 73.94
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.53, 95% CI 2-sided [2.90 to 7.07]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.01, 95% CI 2-sided [2.36 to 6.80]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.23, 95% CI 2-sided [2.82 to 9.72]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.25, 95% CI 2-sided [2.63 to 10.47]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 6.53, 95% CI 2-sided [3.16 to 13.48]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 8.38, 95% CI 2-sided [3.86 to 18.17]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.84, 95% CI 2-sided [3.94 to 15.62]

35. Secondary Outcome: Percentage of Participants Achieving DAS28 Improvement of ≥0.6 From Baseline at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 30
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 97.31 | 96.03
  Week 50 (N: 260, 126) | 98.46 | 97.62
  Week 63 (N: 260, 126) | 96.92 | 99.21
  Week 76 (N: 260, 126) | 96.54 | 99.21
  Week 89 (N: 241, 120) | 96.27 | 99.17
  Week 102 (N: 241, 120) | 97.10 | 97.50
  Week 115 (N: 241, 120) | 97.10 | 95.00
  Week 128 (N: 241, 120) | 96.68 | 98.33

36. Secondary Outcome: Percentage of Participants Achieving DAS28 Improvement of ≥1.2 From Baseline at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: as for outcome 30
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
percentage of participants
  Week 2 (N: 275, 139) | 57.09 | 26.62
  Week 4 (N: 278, 142) | 78.78 | 44.37
  Week 8 (N: 279, 142) | 87.46 | 58.45
  Week 12 (N: 279, 142) | 89.96 | 62.68
  Week 16 (N: 279, 142) | 92.47 | 68.31
  Week 20 (N: 279, 142) | 93.55 | 64.79
  Week 24 (N: 279, 142) | 90.32 | 61.97
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 3.67, 95% CI 2-sided [2.35 to 5.73]
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.65, 95% CI 2-sided [3.00 to 7.22]
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 4.96, 95% CI 2-sided [3.05 to 8.06]
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.34, 95% CI 2-sided [3.18 to 8.96]
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.70, 95% CI 2-sided [3.23 to 10.06]
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 7.88, 95% CI 2-sided [4.37 to 14.20]
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; Fisher's exact test was used to calculate the p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons; Odds Ratio (OR) = 5.73, 95% CI 2-sided [3.40 to 9.65]

37. Secondary Outcome: Percentage of Participants Achieving DAS28 Improvement of ≥1.2 From Baseline at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 30
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
percentage of participants
  Week 37 (N: 260, 126) | 95.00 | 91.27
  Week 50 (N: 260, 126) | 95.38 | 94.44
  Week 63 (N: 260, 126) | 95.77 | 96.03
  Week 76 (N: 260, 126) | 94.62 | 92.86
  Week 89 (N: 241, 120) | 94.61 | 95.00
  Week 102 (N: 241, 120) | 94.61 | 94.17
  Week 115 (N: 241, 120) | 95.02 | 92.50
  Week 128 (N: 241, 120) | 92.95 | 95.00

38. Secondary Outcome: Change From Baseline in Painful Joint Counts at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: Painful joint count is a physical assessment of the ACR-specified 68 joint set for tenderness/pain. Each joint is rated as either painful or not painful with the total number of painful joints reported as the score. Score range is from 0-68 with lower scores indicating the better outcome.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 2 (N: 278, 140) | -10.28 (0.71) | -5.65 (0.91)
  Week 4 (N: 279, 142) | -15.01 (0.68) | -9.99 (0.87)
  Week 8 (N: 279, 142) | -17.47 (0.63) | -12.27 (0.80)
  Week 12 (N: 279, 142) | -18.70 (0.63) | -13.82 (0.81)
  Week 16 (N: 279, 142) | -19.44 (0.66) | -14.00 (0.85)
  Week 20 (N: 279, 142) | -20.06 (0.62) | -13.85 (0.79)
  Week 24 (N: 279, 142) | -19.77 (0.64) | -12.83 (0.82)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

39. Secondary Outcome: Change From Baseline in Painful Joint Counts at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 38
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 37 (N: 260, 126) | -21.14 (11.76) | -21.43 (13.65)
  Week 50 (N: 260, 126) | -21.47 (11.75) | -22.50 (12.75)
  Week 63 (N: 260, 126) | -21.43 (11.91) | -23.72 (12.74)
  Week 76 (N: 260, 126) | -21.10 (12.42) | -22.90 (12.78)
  Week 89 (N: 241, 120) | -21.55 (11.93) | -23.02 (12.87)
  Week 102 (N: 241, 120) | -21.67 (11.91) | -23.51 (13.13)
  Week 115 (N: 241, 120) | -21.74 (11.82) | -22.72 (12.94)
  Week 128 (N: 241, 120) | -21.44 (12.13) | -23.96 (13.25)

40. Secondary Outcome: Change From Baseline in Swollen Joint Counts at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: Swollen joint count is a physical assessment of the ACR-specified 66 joint set for swelling. Each joint is rated as either swollen or not swollen with the total number of swollen joints reported as the score. Score range is from 0-66 with lower scores indicating the better outcome.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 2 (N: 278, 140) | -7.11 (0.56) | -3.15 (0.72)
  Week 4 (N: 279, 142) | -10.69 (0.49) | -6.98 (0.63)
  Week 8 (N: 279, 142) | -12.96 (0.46) | -8.23 (0.59)
  Week 12 (N: 279, 142) | -14.07 (0.43) | -9.42 (0.56)
  Week 16 (N: 279, 142) | -14.57 (0.40) | -9.78 (0.52)
  Week 20 (N: 279, 142) | -15.21 (0.40) | -9.57 (0.51)
  Week 24 (N: 279, 142) | -15.07 (0.42) | -8.62 (0.55)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

41. Secondary Outcome: Change From Baseline in Swollen Joint Counts at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 40
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 37 (N: 260, 126) | -16.16 (8.75) | -16.01 (10.30)
  Week 50 (N: 260, 126) | -16.54 (8.74) | -17.40 (9.57)
  Week 63 (N: 260, 126) | -16.48 (8.46) | -18.02 (10.27)
  Week 76 (N: 260, 126) | -16.57 (9.02) | -17.71 (10.32)
  Week 89 (N: 241, 120) | -16.69 (8.77) | -18.03 (10.64)
  Week 102 (N: 241, 120) | -16.93 (8.60) | -18.22 (10.84)
  Week 115 (N: 241, 120) | -17.07 (8.71) | -17.76 (11.71)
  Week 128 (N: 241, 120) | -16.58 (8.99) | -18.45 (11.17)

42. Secondary Outcome: Change From Baseline in Physician Global Assessment Score at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: The participant's global disease activity was estimated over the preceding 2-3 days on a scale from 0 (no disease activity) to 10 (extreme disease activity) by the physician.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 2 (N: 278, 140) | -2.68 (0.12) | -1.38 (0.15)
  Week 4 (N: 279, 142) | -3.69 (0.12) | -2.21 (0.16)
  Week 8 (N: 279, 142) | -4.14 (0.12) | -2.63 (0.15)
  Week 12 (N: 279, 142) | -4.25 (0.13) | -2.67 (0.17)
  Week 16 (N: 279, 142) | -4.49 (0.13) | -2.84 (0.16)
  Week 20 (N: 279, 142) | -4.64 (0.12) | -2.85 (0.16)
  Week 24 (N: 279, 142) | -4.75 (0.13) | -2.44 (0.17)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

43. Secondary Outcome: Change From Baseline in Physician Global Assessment Score at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 42
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 37 (N: 260, 126) | -5.03 (1.96) | -4.42 (1.99)
  Week 50 (N: 260, 126) | -5.14 (1.91) | -4.79 (2.09)
  Week 63 (N: 260, 126) | -5.08 (1.97) | -5.02 (1.84)
  Week 76 (N: 260, 126) | -5.18 (1.98) | -4.97 (1.82)
  Week 89 (N: 241, 120) | -5.25 (2.01) | -5.13 (2.09)
  Week 102 (N: 241, 120) | -5.16 (1.87) | -5.18 (1.92)
  Week 115 (N: 241, 120) | -5.26 (1.86) | -5.01 (2.05)
  Week 128 (N: 241, 120) | -5.22 (2.08) | -5.18 (2.00)

44. Secondary Outcome: Change From Baseline in Subject Global Assessment Score at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Description: The participant assessed overall arthritis activity on a scale from 0 (no disease activity) to 10 (extreme disease activity).
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 2 (N: 278, 140) | -2.14 (0.14) | -1.01 (0.18)
  Week 4 (N: 279, 142) | -2.69 (0.15) | -1.54 (0.19)
  Week 8 (N: 279, 142) | -3.13 (0.16) | -1.93 (0.20)
  Week 12 (N: 279, 142) | -3.35 (0.16) | -2.20 (0.21)
  Week 16 (N: 279, 142) | -3.55 (0.16) | -2.33 (0.21)
  Week 20 (N: 279, 142) | -3.83 (0.15) | -2.34 (0.20)
  Week 24 (N: 279, 142) | -3.87 (0.16) | -2.31 (0.21)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

45. Secondary Outcome: Change From Baseline in Subject Global Assessment Score at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 44
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 37 (N: 260, 126) | -3.80 (2.90) | -3.27 (3.16)
  Week 50 (N: 260, 126) | -3.85 (2.82) | -3.44 (2.90)
  Week 63 (N: 260, 126) | -3.83 (2.87) | -3.72 (3.07)
  Week 76 (N: 260, 126) | -3.88 (2.96) | -3.42 (2.80)
  Week 89 (N: 241, 120) | -4.09 (2.92) | -3.91 (2.93)
  Week 102 (N: 241, 120) | -4.14 (2.60) | -3.83 (2.92)
  Week 115 (N: 241, 120) | -4.11 (2.85) | -3.71 (3.11)
  Week 128 (N: 241, 120) | -4.28 (2.73) | -3.82 (2.80)

46. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: The duration of morning stiffness was determined over the preceding 2 days using a 2-question worksheet.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: min
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
min
  Week 2 (N: 276, 137) | -60.59 (8.31) | -11.17 (10.71)
  Week 4 (N: 279, 141) | -74.79 (7.95) | -35.63 (10.21)
  Week 8 (N: 279, 141) | -96.13 (7.84) | -58.55 (10.06)
  Week 12 (N: 279, 141) | -100.2 (7.32) | -64.29 (9.39)
  Week 16 (N: 279, 141) | -96.77 (8.13) | -55.90 (10.44)
  Week 20 (N: 279, 141) | -103.3 (7.30) | -58.21 (9.37)
  Week 24 (N: 279, 141) | -102.1 (8.08) | -53.66 (10.37)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 4; Test type: Superiority or Other; p = 0.0007, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 8; Test type: Superiority or Other; p = 0.0009, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p = 0.0007, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 16; Test type: Superiority or Other; p = 0.0005, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

47. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: The duration of morning stiffness was determined over the preceding 2 days using a 2-question worksheet.
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
min
  Week 37 (N: 260, 125) | -105.39 (189.12) | -87.89 (162.76)
  Week 50 (N: 260, 125) | -105.75 (199.90) | -97.61 (164.68)
  Week 63 (N: 260, 125) | -104.18 (201.17) | -89.61 (170.16)
  Week 76 (N: 260, 125) | -98.83 (202.56) | -91.53 (181.67)
  Week 89 (N: 241, 120) | -125.07 (262.93) | -76.49 (226.83)
  Week 102 (N: 241, 120) | -132.32 (243.81) | -84.53 (205.70)
  Week 115 (N: 241, 120) | -130.55 (267.87) | -89.53 (196.35)
  Week 128 (N: 241, 120) | -118.79 (294.73) | -90.88 (206.55)

48. Secondary Outcome: Change From Baseline in General Health VAS at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: The participants had to indicate on a 100 mm-VAS (0 mm: very well, 100 mm: extremely bad) in general how they rated their health over the preceding 2-3 weeks.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
mm
  Week 2 (N: 278, 140) | -20.51 (1.43) | -8.75 (1.82)
  Week 4 (N: 279, 142) | -25.23 (1.49) | -13.11 (1.90)
  Week 8 (N: 279, 142) | -28.17 (1.60) | -17.00 (2.04)
  Week 12 (N: 279, 142) | -30.54 (1.57) | -19.60 (2.00)
  Week 16 (N: 279, 142) | -32.69 (1.66) | -21.04 (2.11)
  Week 20 (N: 279, 142) | -34.69 (1.50) | -20.04 (1.91)
  Week 24 (N: 279, 142) | -33.71 (1.58) | -19.27 (2.01)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

49. Secondary Outcome: Change From Baseline in General Health VAS at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 48
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
mm
  Week 37 (N: 260, 126) | -34.48 (29.60) | -31.02 (29.91)
  Week 50 (N: 260, 126) | -33.47 (27.53) | -31.51 (25.99)
  Week 63 (N: 260, 126) | -33.53 (28.05) | -34.33 (27.40)
  Week 76 (N: 260, 126) | -33.25 (28.44) | -33.11 (27.12)
  Week 89 (N: 241, 120) | -34.79 (29.13) | -34.78 (26.96)
  Week 102 (N: 241, 120) | -34.84 (27.07) | -35.30 (27.60)
  Week 115 (N: 241, 120) | -34.86 (27.41) | -32.11 (27.75)
  Week 128 (N: 241, 120) | -36.25 (27.09) | -36.35 (27.57)

50. Secondary Outcome: Change From Baseline in Pain VAS at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: The participants had to indicate on a 100 mm-VAS (0 mm: no pain, 100 mm: pain as bad as it could be) the amount of pain they experienced over the preceding 2-3 days.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
mm
  Week 2 (N: 278, 140) | -27.66 (1.48) | -10.46 (1.90)
  Week 4 (N: 279, 142) | -31.58 (1.60) | -16.30 (2.04)
  Week 8 (N: 279, 142) | -36.05 (1.60) | -23.45 (2.05)
  Week 12 (N: 279, 142) | -37.24 (1.65) | -23.74 (2.11)
  Week 16 (N: 279, 142) | -39.86 (1.62) | -24.30 (2.07)
  Week 20 (N: 279, 142) | -40.59 (1.57) | -24.75 (2.01)
  Week 24 (N: 279, 142) | -40.91 (1.62) | -23.97 (2.08)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

51. Secondary Outcome: Change From Baseline in Pain VAS at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 50
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
mm
  Week 37 (N: 260, 126) | -41.66 (27.84) | -36.89 (29.64)
  Week 50 (N: 260, 126) | -40.49 (27.84) | -36.63 (27.71)
  Week 63 (N: 260, 126) | -39.98 (27.23) | -39.36 (26.85)
  Week 76 (N: 260, 126) | -40.38 (28.94) | -37.17 (27.12)
  Week 89 (N: 241, 120) | -42.37 (29.14) | -38.55 (28.17)
  Week 102 (N: 241, 120) | -41.99 (27.73) | -39.85 (27.69)
  Week 115 (N: 241, 120) | -42.27 (26.65) | -36.92 (27.55)
  Week 128 (N: 241, 120) | -41.95 (28.56) | -40.57 (26.81)

52. Secondary Outcome: Change From Baseline in Fatigue VAS at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: The participants had to indicate on a 100 mm-VAS (0 mm: no fatigue, 100 mm: a great deal of fatigue) how much of a problem had fatigue or tiredness been for them in the preceding week.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
mm
  Week 2 (N: 278, 140) | -18.64 (1.48) | -6.29 (1.90)
  Week 4 (N: 279, 142) | -21.54 (1.59) | -10.44 (2.04)
  Week 8 (N: 279, 142) | -26.66 (1.55) | -16.04 (1.98)
  Week 12 (N: 279, 142) | -27.40 (1.63) | -16.45 (2.08)
  Week 16 (N: 279, 142) | -29.10 (1.68) | -16.87 (2.15)
  Week 20 (N: 279, 142) | -30.74 (1.61) | -18.95 (2.06)
  Week 24 (N: 279, 142) | -29.57 (1.64) | -17.26 (2.10)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

53. Secondary Outcome: Change From Baseline in Fatigue VAS at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 52
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
mm
  Week 37 (N: 260, 126) | -30.76 (29.09) | -23.69 (29.10)
  Week 50 (N: 260, 126) | -29.03 (31.59) | -25.32 (30.94)
  Week 63 (N: 260, 126) | -28.95 (31.51) | -28.74 (31.19)
  Week 76 (N: 260, 126) | -29.44 (31.48) | -28.17 (28.16)
  Week 89 (N: 241, 120) | -30.75 (30.78) | -28.38 (31.05)
  Week 102 (N: 241, 120) | -30.37 (31.42) | -30.61 (30.08)
  Week 115 (N: 241, 120) | -30.87 (30.83) | -27.38 (29.51)
  Week 128 (N: 241, 120) | -30.52 (31.26) | -30.35 (30.65)

54. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score Using vdH mTSS at Week 24
Description: mTSS: sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Each x-ray visit included 4 films, each of which were read by 2 readers. The mTSS was calculated by the images scored for erosions and JSN. An increase in mTSS from Baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Week 24
Population: xITT population included all participants who took at least 1 dose of study drug and had evaluable radiographic data at Baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 247 | 119
units on a scale | -0.01 (0.22) | 0.23 (0.28)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-value; Test type: Superiority or Other; p = 0.1975, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

55. Secondary Outcome: Change From Baseline in Erosion Score Using vdH mTSS at Week 24
Description: as for outcome 54
Time Frame: Week 24
Population: as for outcome 54
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 247 | 119
units on a scale | 0.42 (0.22) | 1.14 (0.29)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 54, analysis 1]; Test type: Superiority or Other; p = 0.0044, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

56. Secondary Outcome: Change From Baseline in Westergren ESR at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hour. A higher rate is consistent with inflammation. ESR was performed at the investigative site using an ESR kit supplied by the centralized laboratory.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm/hour
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
mm/hour
  Week 2 (N: 275, 139) | -13.16 (0.96) | -4.35 (1.24)
  Week 4 (N: 278, 142) | -17.31 (0.99) | -8.06 (1.27)
  Week 8 (N: 279, 142) | -18.68 (1.03) | -10.11 (1.31)
  Week 12 (N: 279, 142) | -19.74 (1.11) | -12.53 (1.42)
  Week 16 (N: 279, 142) | -20.48 (1.07) | -12.87 (1.37)
  Week 20 (N: 279, 142) | -20.56 (1.12) | -12.60 (1.44)
  Week 24 (N: 279, 142) | -20.72 (1.16) | -12.37 (1.48)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

57. Secondary Outcome: Change From Baseline in Westergren ESR at Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Description: as for outcome 56
Time Frame: Week 37, Week 50, Week 63, Week 76, Week 89, Week 102, Week 115, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
mm/hour
  Week 37 (N: 260, 126) | -19.56 (18.40) | -20.25 (14.92)
  Week 50 (N: 260, 126) | -18.48 (19.62) | -20.27 (16.78)
  Week 63 (N: 260, 126) | -18.26 (18.56) | -18.31 (17.68)
  Week 76 (N: 260, 126) | -17.78 (18.74) | -17.54 (20.00)
  Week 89 (N: 241, 120) | -18.23 (19.04) | -17.08 (19.74)
  Week 102 (N: 241, 120) | -15.20 (20.32) | -16.63 (19.00)
  Week 115 (N: 241, 120) | -15.65 (19.83) | -15.30 (21.70)
  Week 128 (N: 241, 120) | -13.75 (22.36) | -15.48 (20.59)

58. Secondary Outcome: Change From Baseline in CRP at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. CRP was analysed at a central laboratory.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
mg / dL
  Week 2 (N: 277, 139) | -13.39 (1.30) | -0.62 (1.66)
  Week 4 (N: 279, 142) | -11.88 (1.28) | -3.15 (1.64)
  Week 8 (N: 279, 142) | -11.81 (1.36) | -4.52 (1.74)
  Week 12 (N: 279, 142) | -12.33 (1.34) | -5.80 (1.72)
  Week 16 (N: 279, 142) | -12.98 (1.31) | -5.81 (1.67)
  Week 20 (N: 279, 142) | -12.32 (1.18) | -4.39 (1.52)
  Week 24 (N: 279, 142) | -12.31 (1.18) | -7.06 (1.51)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 4]; Test type: Superiority or Other; p = 0.0007, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 6]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 7: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p = 0.0021, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

59. Secondary Outcome: Change From Baseline in SF-36 Health Survey Vitality Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 3.43 (0.26) | 2.00 (0.33)
  Week 16 (N: 278, 138) | 3.90 (0.26) | 2.37 (0.34)
  Week 24 (N: 278, 138) | 3.79 (0.27) | 2.36 (0.35)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

60. Secondary Outcome: Change From Baseline in SF-36 Health Survey Vitality Domain Score at Week 50, Week 76, Week 102, and Week 128
Description: as for outcome 3
Time Frame: Week 50, Week 76, Week 102, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 50 (N: 259, 126) | 4.08 (4.72) | 3.56 (4.04)
  Week 76 (N: 259, 126) | 3.71 (4.83) | 3.49 (4.16)
  Week 102 (N: 241, 120) | 4.00 (4.55) | 3.60 (4.64)
  Week 128 (N: 241, 120) | 3.89 (4.95) | 3.62 (4.28)

61. Secondary Outcome: Change From Baseline in SF-36 Health Survey Mental Component Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 6.85 (0.65) | 2.98 (0.84)
  Week 16 (N: 278, 138) | 6.70 (0.68) | 4.51 (0.87)
  Week 24 (N: 278, 138) | 7.33 (0.73) | 3.32 (0.95)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0264, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

62. Secondary Outcome: Change From Baseline in SF-36 Health Survey Mental Component Score at Week 50, Week 76, Week 102, and Week 128
Description: as for outcome 3
Time Frame: Week 50, Week 76, Week 102, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 50 (N: 259, 126) | 8.28 (11.62) | 5.61 (9.95)
  Week 76 (N: 259, 126) | 7.39 (12.71) | 6.61 (10.66)
  Week 102 (N: 241, 120) | 7.19 (12.49) | 6.05 (11.61)
  Week 128 (N: 241, 120) | 7.32 (12.86) | 6.42 (11.48)

63. Secondary Outcome: Change From Baseline in SF-36 Health Survey Physical Component Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 10.08 (0.60) | 7.04 (0.78)
  Week 16 (N: 278, 138) | 12.26 (0.63) | 7.98 (0.82)
  Week 24 (N: 278, 138) | 12.44 (0.65) | 7.36 (0.84)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0005, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

64. Secondary Outcome: Change From Baseline in SF-36 Health Survey Physical Component Score at Week 50, Week 76, Week 102, and Week 128
Description: as for outcome 3
Time Frame: Week 50, Week 76, Week 102, and Week 128
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 260 | 126
units on a scale
  Week 50 (N: 259, 126) | 13.07 (10.19) | 12.32 (9.59)
  Week 76 (N: 259, 126) | 12.84 (10.77) | 11.29 (10.37)
  Week 102 (N: 241, 120) | 13.77 (10.17) | 12.28 (9.84)
  Week 128 (N: 241, 120) | 13.47 (10.64) | 12.10 (9.68)

65. Secondary Outcome: Change From Baseline in SF-36 Health Survey Bodily Pain Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 2.93 (0.15) | 1.84 (0.19)
  Week 16 (N: 278, 138) | 3.24 (0.15) | 2.24 (0.20)
  Week 24 (N: 278, 138) | 3.39 (0.16) | 2.00 (0.21)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; ANCOVA model with Baseline as covariate and factors for treatment and country as class variables was used to calculate p-values. ANCOVA was ran at each time-point shown, however as p-values obtained were identical, only one p-value is presented (which is applicable to each time-point - Week 8, Week 16, and Week 24 - independently); Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

66. Secondary Outcome: Change From Baseline in SF-36 Health Survey Role Limitations Due to Emotional Problems Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 0.87 (0.09) | 0.51 (0.11)
  Week 16 (N: 278, 138) | 0.89 (0.09) | 0.66 (0.12)
  Week 24 (N: 278, 138) | 1.04 (0.09) | 0.46 (0.11)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0061, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0730, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

67. Secondary Outcome: Change From Baseline in SF-36 Health Survey General Health Perceptions Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 3.22 (0.25) | 2.25 (0.32)
  Week 16 (N: 278, 138) | 3.62 (0.25) | 2.56 (0.32)
  Week 24 (N: 278, 138) | 3.95 (0.26) | 2.14 (0.34)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0066, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0036, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

68. Secondary Outcome: Change From Baseline in SF-36 Health Survey Mental Health Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 3.21 (0.30) | 1.25 (0.38)
  Week 16 (N: 278, 138) | 3.62 (0.30) | 2.21 (0.39)
  Week 24 (N: 278, 138) | 3.59 (0.33) | 1.81 (0.42)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0013, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

69. Secondary Outcome: Change From Baseline in SF-36 Health Survey Physical Functioning Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 3.97 (0.30) | 2.63 (0.39)
  Week 16 (N: 278, 138) | 4.95 (0.32) | 3.08 (0.41)
  Week 24 (N: 278, 138) | 5.06 (0.33) | 2.86 (0.42)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0021, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

70. Secondary Outcome: Change From Baseline in SF-36 Health Survey Role Limitations Due to Physical Health Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 1.36 (0.12) | 0.88 (0.15)
  Week 16 (N: 278, 138) | 1.67 (0.12) | 1.08 (0.15)
  Week 24 (N: 278, 138) | 1.65 (0.12) | 0.90 (0.15)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p = 0.0062, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0007, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

71. Secondary Outcome: Change From Baseline in SF-36 Health Survey Social Functioning Domain Score at Week 8, Week 16, and Week 24
Description: as for outcome 3
Time Frame: Week 8, Week 16, and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept + Methotrexate | DMARD + Methotrexate
Number analyzed (Participants) | 279 | 142
units on a scale
  Week 8 (N: 278, 138) | 1.51 (0.12) | 0.77 (0.15)
  Week 16 (N: 278, 138) | 1.45 (0.13) | 0.95 (0.16)
  Week 24 (N: 278, 138) | 1.60 (0.12) | 0.82 (016)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 5]; Test type: Superiority or Other; p = 0.0073, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Etanercept + Methotrexate vs DMARD + Methotrexate; [analysis description as in outcome 46, analysis 7]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided, without any adjustment for multiple comparisons

ADVERSE EVENTS:
Time Frame: Phase 1: Baseline-Week 26 (Follow up telephone visit), Phase 2 Year 1: Week 24-Week 76, Phase 2 Year 2: Week 76-Week 128
Description: The same event may appear as both an AE and a SAE. DMARD + methotrexate included 143 rather than 142 participants as reported in the Phase 1 CSR. One participant was originally excluded from evaluation for no record of dosing, however 4 days of study medication was later reported.
Groups:
- Etanercept + Methotrexate Phase 1; Etanercept + Methotrexate Phase 2 Year 1; Etanercept + Methotrexate Phase 2 Year 2: Phase 1: Etanercept 50 mg injection s.c. once weekly along with methotrexate tablet (7.5-25 mg) orally once weekly either in single dose or in 2 divided doses for 24 weeks. Phase 2: During the optional Phase 2-period (week 24-week 128), the participants could remain on etanercept and methotrexate, or a non-biologic DMARD the investigator preferred in accordance with the local label (SSZ or HCQ) could be added in exchange for or in addition to etanercept. Methotrexate could be continued, discontinued or titrated. Phase 1 reporting groups were used also for Phase 2 data, regardless of the participant's Phase 2 treament regimen.
- DMARD + Methotrexate Phase 1; DMARD + Methotrexate Phase 2 Year 1; DMARD + Methotrexate Phase 2 Year 2: Phase 1: Conventional DMARD combination therapy (SSZ or HCQ) tablets administered as per local prescribing practice, along with methotrexate tablet (7.5-25 mg) orally once weekly either in single dose or in 2 divided doses for 24 weeks. Phase 2: During the optional Phase 2-period (week 24-week 128), the participants could remain on DMARD (SSZ or HCQ) and methotrexate, or a DMARD the investigator preferred in accordance with the local label (HCQ, SSZ, and/or etanercept) could be added in exchange for or in addition to the Phase 1 DMARD (SSZ or HCQ). Methotrexate and the DMARD administered in Phase 1 could be continued, discontinued or titrated. Phase 1 reporting groups were used also for Phase 2 data, regardless of the participant's Phase 2 treament regimen.
Arm/Group | Etanercept + Methotrexate Phase 1 | DMARD + Methotrexate Phase 1 | Etanercept + Methotrexate Phase 2 Year 1 | DMARD + Methotrexate Phase 2 Year 1 | Etanercept + Methotrexate Phase 2 Year 2 | DMARD + Methotrexate Phase 2 Year 2
Serious Adverse Events (participants affected / at risk) | 10/281 | 2/143 | 17/260 | 4/126 | 11/241 | 2/120
Other Adverse Events (participants affected / at risk) | 64/281 | 41/143 | 19/260 | 19/126 | 37/241 | 20/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept + Methotrexate Phase 1 (N=281) | DMARD + Methotrexate Phase 1 (N=143) | Etanercept + Methotrexate Phase 2 Year 1 (N=260) | DMARD + Methotrexate Phase 2 Year 1 (N=126) | Etanercept + Methotrexate Phase 2 Year 2 (N=241) | DMARD + Methotrexate Phase 2 Year 2 (N=120)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular vascular disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Borderline serous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept + Methotrexate Phase 1 (N=281) | DMARD + Methotrexate Phase 1 (N=143) | Etanercept + Methotrexate Phase 2 Year 1 (N=260) | DMARD + Methotrexate Phase 2 Year 1 (N=126) | Etanercept + Methotrexate Phase 2 Year 2 (N=241) | DMARD + Methotrexate Phase 2 Year 2 (N=120)
Dyspepsia (Gastrointestinal disorders) | 6 | 9 | 3 | 2 | 3 | 0
Gastritis (Gastrointestinal disorders) | 5 | 9 | 5 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 7 | 13 | 5 | 4 | 4 | 3
Bronchitis (Infections and infestations) | 18 | 3 | 11 | 10 | 17 | 3
Influenza (Infections and infestations) | 15 | 6 | 11 | 4 | 9 | 6
Nasopharyngitis (Infections and infestations) | 14 | 5 | 11 | 11 | 11 | 4
Urinary tract infection (Infections and infestations) | 8 | 5 | 10 | 5 | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 5 | 1 | 3 | 6
Headache (Nervous system disorders) | 11 | 10 | 7 | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.